CLINICAL TRIAL: NCT00615823
Title: Clinical Effect and Tolerability of Atorvastatin Versus Placebo in Patients With Pulmonary Hypertension: Double-blinded, Randomised, Prospective Phase II Study for 6 Months With Adjusted Doses of Atorvastatin
Brief Title: Atorvastatin in Pulmonary Hypertension
Acronym: APATH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: National Grant from The Ministry of Science and Technology (Unknown); Capital Development Scientific Fund (Unknown)
Responsible Party: Principal Investigator, Jianguo He, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-1152; 2006BAI01A07 (Other Grant/Funding Number: National Grant from The Ministry of Science); 2005-1018 (Other Grant/Funding Number: Capital Development Scientific Fund)
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Atorvastatin group: receive atorvastatin 10 mg daily in addition to supportive care
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Placebo group: receive matching placebo in addition to supportive care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Patients were assigned to receive 10 mg of atorvastatin for 6 months (supplied by JiaLin Pharmaceutical Co., Beijing, China). The dose was adjusted to 5mg daily if serum transaminase levels increased by less than three times the upper limit of normal or creatine kinase levels increased to less than five times the upper limit of normal. If serum transaminase and creatine kinase levels remained normal and low-density lipoprotein level greater than 3.4mmol/L after 4 weeks of therapy, the dose of drug was increased to 20mg once daily.
  Other Names: atorvastatin: a'le(bland names)
  Arms: 1
Drug: Placebo — Patients were assigned to receive 10 mg of placebo for 6 months (supplied by JiaLin Pharmaceutical Co., Beijing, China). The dose was adjusted to 5mg daily if serum transaminase levels increased by less than three times the upper limit of normal or creatine kinase levels increased to less than five times the upper limit of normal. If serum transaminase and creatine kinase levels remained normal and low-density lipoprotein level greater than 3.4mmol/L after 4 weeks of therapy, the dose of drug was increased to 20mg once daily.
  Other Names: matching placebo: a'le(brand name)
  Arms: 2

SUMMARY:
Clinical effect and tolerability of atorvastatin versus placebo in patients with Pulmonary Hypertension: double-blinded, randomised, prospective phase II study for 6 months with adjusted doses of Atorvastatin

DETAILED DESCRIPTION:
PAH is characterized by dyspnea, fatigue, and lower extremity edema as a result of heart failure. Several research have proved that inflammation may participate in the pathogenesis of PAH. As atorvastatin inhibits inflammation and has beneficial effects on blood vessels in other types of cardiovascular disease. Therefore, atorvastatin may similarly benefit patients with PAH. Experimental data suggest that statins attenuates pulmonary hypertension in animal experiments. In addition, non-controlled clinical studies suggest that atorvastatin is effective and safe in patients with pulmonary hypertension.

Participants in this study will be randomly assigned to receive 6 months of daily placebo tablets or daily atorvastatin in a double-blind fashion. The study will compare the safety and efficacy of placebo and atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign the informed consent form
* <=65 and >=18years old
* Diagnosis of pulmonary arterial hypertension (Mean pulmonary artery pressure greater than 25 mm Hg at rest with a pulmonary capillary wedge pressure less than 15 mm Hg )that is a) idiopathic, b) familial, or c) associated with connective-tissue disease, d)congenital systemic-to-pulmonary shunt occurring after surgical/interventional repair that had been performed at least five years previously or in the absence of indications for surgery/intervention treatment e) chronic thromboembolism PAH in the absence of indications for surgery
* Patients in WHO functional class II to III
* Vasodilator Testing nonresponders
* Baseline six-minute walking distance between 100 and 460 m

Exclusion Criteria:

* PAH related to other etiologies (Groups 2, 3 and 5 pulmonary hypertension)
* A forced expiratory volume in one second/ forced vital capacity bellow 50% or a total lung capacity of less than 60 percent predicted value
* A 6-minute walk distance of less than 100 or more than 460 m
* A positive acute vasodilator response
* Current treatment with calcium-channel blockers or specific therapy (endothelin receptor antagonist, phosphodiesterase-5 inhibitor, or prostacyclin)
* Inability to perform 6-minute walk test
* Serum transaminase level three times above the upper limit of normal
* Creatine kinase level five times above the upper limit of normal
* Previously diagnosed heart disease such as serious cardiac arrhythmias, unstable angina pectoris, myocardial infarction
* History of transient ischemia attack or stroke within three months
* Bleeding disorder
* Positive pregnancy test or breastfeeding practice
* History or suspicion of inability to cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-02; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The placebo-corrected change from baseline to week 24 in 6-minute walk distance | Measured at 6 months

SECONDARY OUTCOMES:
Time from randomization to clinical worsening | Measured at 6 months
  Clinical worsening was defined as death, the first occurrence of hospitalization for pulmonary arterial hypertension, or initiation of PAH-specific drug therapy
Change from baseline to week 24 in World Health Organization functional class | measured at 6 monthes
  World Health Organization (WHO) functional class: an adaptation of the New York Heart Association classification.
Change from baseline to week 24 in Borg dyspnea score | measured at 6 monthes
  Borg dyspnea score: with 0 representing no dyspnea and 10 maximal dyspnea.
Change from baseline to week 24 in hemodynamic parameters derived from right heart catheterization. | measured at 6 monthes
  Hemodynamic parameters: mean pulmonary artery pressure, right atrial pressure, cardiac index and pulmonary vascular resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo He, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Cardiovascular Institute and Fu Wai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zeng WJ, Xiong CM, Zhao L, Shan GL, Liu ZH, Xue F, Gu Q, Ni XH, Zhao ZH, Cheng XS, Wilkins MR, He JG; Atorvastatin in Pulmonary Arterial Hypertension (APATH) Study Group. Atorvastatin in pulmonary arterial hypertension (APATH) study. Eur Respir J. 2012 Jul;40(1):67-74. doi: 10.1183/09031936.00149011. Epub 2012 Feb 23. PMID 22362846